CLINICAL TRIAL: NCT05694052
Title: Impact of the Use a Multifaceted Intervention of Environment Control in the ICU to Optimize Quantity and Quality of Sleep in Critically Ill Patients
Brief Title: Impact of a Multifaceted Intervention of Environment Control in the ICU to Optimize Quantity and Quality of Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Agencia Nacional de Investigacion y Desarrollo, ANID (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 190528002; 1201772 (Other: FONDECYT)
Record Dates: First submitted 2022-06-30; First posted 2023-01-23 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-08

CONDITIONS: Sleep Disturbance
Keywords: ICU; Environment control; Critically ill patients; Adult; Multifaceted intervention
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: Prospective, parallel-group, randomized trial in critically ill patients. The project will follow the CONSORT guidelines for this class of studies.
  Patients randomized sequence will be generated by a computer program with an allocation 1:1. They will be randomized to receive a multifaceted intervention of environmental control in the ICU (intervention group) or standard care (control group).
Who Masked: Outcomes Assessor
Masking Description: Due to the type of intervention under study, the patient and the research team can not be blinded to the group assignment. Statisticians and the researchers responsible for analysis of PSG and actigraphy, as well as those performing long-term outcome assessments, will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multifaceted Intervention (Experimental): Lighting: a multi-channel LED Spectrum will be implemented. The spectral output covers the wavelength range from 420 nm to 730 nm. All active channels are mixed, providing a smooth (uniform in color) light with a Lambertian pattern profile.
  Noise: the auditory masking system will provide a continuous background digitally generated broadband pink noise. The sound system will be placed near the head of the bed. This will be started (at 62 DB sound level) each night for 8 hours.
  Nocturnal patient care activities: night-time patient care activities will be re-organized to minimize interruptions. The medication administration schedule will be organized, and the vital signs monitoring will be done continuously by medical devices without requiring to disturb the patient. Hygiene, comfort, and elective activities will be scheduled for the daytime. Emergency interventions will not be limited.
  Interventions: Behavioral: Multifaceted Intervention of environment control
- Standard Care (No Intervention): Lighting: standard lighting system currently installed in the ICU rooms provides a fix light of 300 to 400 lux during daytime, and 0 to 30 lux during night-time. Controls depends on staff to switched on and off.
  Noise: The rooms do not have noise isolation and there is no protocol for reducing environmental noise. In our ICU, isolated measurements reported mean average values of 60 dB during daytime and 50 dB during nighttime, with frequent peaks over 80 to 90 dB.
  Nocturnal patient care activities: There is no specific protocol for patient care activities during the night. The activities (schedules of drug administration and intravenous infusions, non-urgent examinations, and non-urgent procedures) are organized during the morning by the patient's nurse according to their own clinical criteria. Hygiene and comfort activities are carried out in standard schedules according to the rules of the ICU. Drug administration, examinations and urgent procedures are performed when necessary.

INTERVENTIONS:
Behavioral: Multifaceted Intervention of environment control — Dynamic light therapy, auditory masking, and rationalization of ICU nocturnal patient activities.
  Arms: Multifaceted Intervention

SUMMARY:
In critically ill patients, sleep and circadian rhythms are markedly disturbed, including sleep deprivation and disruption, as well as altered sleep architecture, and loss of normal oscillations of Melatonin and Cortisol. These alterations have been associated with delirium, fatigue, and higher mortality. In addition, sleep disturbances may remain after hospital discharge, and they have been associated with psychological comorbidities, which may contribute to the low quality of life observed in ICU survivors. Patient factors for sleep deprivation in ICU are the type/severity of underlying illness, the pathophysiology of the acute illness, pain, and stress/anxiety. Factors associated with the ICU, such as exposure to inadequate levels of light and noise, or inflexible schedules of daily care activities, have also been reported to have a major role in sleep disturbance.

A limited number of studies have evaluated interventions targeting sleep optimization in the ICU, using strategies like eye masks and/or earplugs to isolate patients from their environment, the application of a dynamic light system that ensures light at night and higher levels of light at daytime to restore circadian rhythm, or auditory masking, to avoid intense cortical stimuli secondary to annoying noises. These strategies have been reported to have some positive impacts on sleep in ICU but this has only been assessed by qualitative instruments. In addition, they have been tested as isolated interventions, and not as part of a more comprehensive approach.

The goal of this project is to determine the impact of a multifaceted intervention of environmental control in the ICU, based on dynamic light therapy, auditory masking, and rationalization of ICU nocturnal patient care activities, on quantity and quality of sleep, assessed by polysomnography and other semi-quantitative methods, compared to standard care. In addition, the effect of both strategies on delirium, circadian rhythm biomarkers, and long-term neuropsychological outcomes will be compared.

This is a prospective, parallel-group, randomized trial in 56 critically ill patients once they are starting to recover from their acute illness. After obtaining informed consent, patients will be randomized to receive a multifaceted intervention of environmental control or standard care. And this protocol will be applied from enrollment until ICU discharge, with a follow-up before hospital discharge and at 6 months.

DETAILED DESCRIPTION:
Sleep can be defined as a periodic and reversible state of disengagement from the environment. It consists of an active process that involves multiple, complex physiological and behavioral mechanisms of the central nervous system. It is also a natural process highly conserved during evolution, which is critical for health and well-being, being essential for rest, repair, and for the survival of the individual. Sleep is controlled by a circadian system that drives 24-h periodicity, and a homeostatic system that ensures that adequate amounts of sleep are obtained, and it can be assessed in terms of quantity (total sleep time, and time spent in each sleep stage), quality (fragmentation, sleep stage changes, wake after sleep onset, EEG sleep patterns), and distribution over the 24-h cycle.

The ICU can be a hostile and stressful environment for patients. From the point of view of ICU survivors, a stay in the critical care unit represents a traumatic event in their lives and the environment does not favor rest, due to the equipment (alarms from monitors and life-supporting devices) and human factors (staff conversations), all related to therapy and care.

In critically ill patients, sleep and circadian rhythms are markedly disturbed. Abnormalities include sleep deprivation and disruption, as well as altered sleep architecture, and loss of normal oscillations of melatonin and cortisol. These alterations have been associated with delirium, fatigue, and higher mortality. In addition, sleep disturbances may remain after hospital discharge and have been consistently associated with psychological comorbidities, which may contribute to the low quality of life observed in ICU survivors. Patient factors for sleep deprivation in ICU are the type and severity of the underlying illness, the pathophysiology of the acute illness, pain (from procedures or the underlying condition), and stress/anxiety. Most of these factors are intrinsic to ICU patients and therefore, difficult to modify. However, factors associated with the ICU environment, such as exposure to inadequate levels of light and noise during the day and night, or inflexible schedules of daily care activities, have also been reported to have a major role in sleep disturbance. For decades these aspects of ICU care had received little attention but in recent years there has been increasing interest in changing this reality.

A limited number of studies have evaluated interventions targeting sleep optimization in the ICU. The most studied strategy to date has been the use of eye masks and/or earplugs, however, studies report poor tolerance for them. A more complex but interesting intervention to restore circadian rhythm is the application of a dynamic light system, that ensures low light at night and higher levels of light at the daytime. In terms of noise, an interesting alternative is to apply auditory masking to avoid intense cortical stimuli secondary to annoying noises, and therefore prevent awakenings. These strategies have been reported to have some positive impacts on sleep in ICU, but sleep has only been assessed by qualitative methods. In addition, they have been tested as isolated interventions, and not as part of a more comprehensive approach.

A proposal is an interdisciplinary approach, which targets different environmental factors and integrates experts from different fields. Although the concepts of dynamic light and sound masking are well known, our proposal includes the local design of solutions based on these concepts. This study also chose to use the highest standard for sleep measurements (PSG), which has been one of the main limitations of previous research in this field. It is hoped that the intervention will be effective in improving sleep. Although this study is underpowered to study the potential impacts of the strategy on mortality or ICU length of stay, if the intervention proves to be effective in improving sleep, a larger-scale study could follow. But even if the intervention proves not to be effective, the data collected about sleep and about long-term neuropsychological outcomes in our ICU population will be highly relevant to advance our understanding of the relation between these variables, and for the planning of future studies.

The hypothesis is that the use of a multifaceted intervention of environmental control in the ICU, based on dynamic light therapy, auditory masking, and rationalization of ICU nocturnal patient care activities, is associated with improved quantity and quality of sleep, assessed by polysomnography and other semiquantitative methods, compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patient under invasive mechanical ventilation for at least 72 hours.
* Patient without sedation or with superficial sedation level (SAS 3-4 by Sedation- Agitation Scale), during most of the daytime within the 24 previous hours

Exclusion Criteria:

* Patient who required mechanical ventilation in another episode of hospitalization in the 2 months before screening.
* Patients with primary neurological or neurosurgical disease.
* Presence of mental or intellectual disability prior to hospitalization or communication/language barriers.
* Pre-existing comorbidity with a life expectancy not exceeding 6 months (eg, metastatic cancer).
* Readmission to the ICU (patients can only be included if they are on their first ICU admission of the present hospitalization).
* No fixed address for follow-up.
* Patients with moderate to severe visual or hearing impairment.
* Patients with known sleep disturbance before hospital admission.
* Early limitation of therapeutic effort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Minutes in slow-wave sleep-N3 | Night 3 from enrollment.
  Minutes in slow-wave sleep-N3 evaluated by Polysomnography.

SECONDARY OUTCOMES:
Minutes of rapid eye movement sleep | Night 3 from enrollment.
  Minutes of rapid eye movement sleep evaluated by Polysomnography.
Total sleep time | From the first day after randomization, assessed up 1 week after ICU discharge.
  Assessed by actigraphy. It will report the total sleep duration in minutes within each 24-hour period.
Change in Richards-Campbell Sleep Questionnaire (RCSQ) score | From the second day of enrollment until discharge from ICU, assessed up to day 28.
  The Richards-Campbell Sleep Questionnaire (RCSQ) is a 5-item questionnaire used to evaluate perceived sleep depth, sleep latency, number of awakenings, efficiency, and sleep quality. Each RCSQ question is measured on a 0 (minimum) to 100 (maximum) visual-analog scale, with higher scores representing better sleep.
Change in Pittsburgh Sleep Quality Index (PSQI) score | From the second day of enrollment until discharge from ICU, assessed up to day 28.
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measure seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Circadian rhythm | Melatonin and cortisol plasmatic levels will be assessed at the day 1 and 3 after randomization.
  Oscillation of plasma concentration of melatonin and cortisol will be assessed. Five samples will be taken each day.
Incidence of Delirium in ICU | From the first day of enrollment after randomization and until ICU discharge, assessed up to day 28.
  The incidence of delirium is monitored and evaluated by the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). The CAM-ICU has four items ((1) altered mental status/fluctuating course, (2)inattention, (3) altered level of consciousness, and (4) disorganized thinking) and each item has two factors (positive or negative). The physicians can diagnose the patients with delirium when the results of item (1), item (2), and item (3) or item (4) are positive.
Duration of delirium (in days) | From the first day of enrollment after randomization and until ICU discharge, assessed up to day 28.
  Evaluated by Confusion Assessment Method for the ICU (CAM-ICU). Duration of delirium will be defined as the total days of delirium during ICU stay.
Hospital Anxiety and Depression Scale (HADS) | 6 months post ICU discharge
  The HADS is a 14-item(1 - 4 points) measure designed to assess anxiety and depression symptoms in medical patients. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D). Scores higher than 11 on either scale indicate a definitive case.
Global cognition as measured by Montreal Cognitive Assessment (MOCA) | 6 months post ICU discharge.
  Measured by the Montreal Cognitive Assessment (MOCA, minimum score 0 maximum score 30, with higher scores suggesting better cognitive performance)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro R Bruhn, PhD, Study Chair — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clínico UC CHRISTUS, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Alegria L, Brockmann P, Repetto P, Leonard D, Cadiz R, Paredes F, Rojas I, Moya A, Oviedo V, Garcia P, Bakker J. Improve sleep in critically ill patients: Study protocol for a randomized controlled trial for a multi-component intervention of environment control in the ICU. PLoS One. 2023 May 25;18(5):e0286180. doi: 10.1371/journal.pone.0286180. eCollection 2023. PMID 37228142